CLINICAL TRIAL: NCT04113915
Title: Viral Hepatitis B and C Infection in Patients With Idiopathic Thrombocytopenic Purpura Treated With Triple Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Safaa AA Khaled (Other)
Responsible Party: Sponsor-Investigator, Safaa AA Khaled, Assisstant professor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Viral hepatitis in ITP
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: ITP - Immune Thrombocytopenic Purpura; Viral Hepatitis
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Cyclosporine; Rituximab; Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group of ITP patients received triple therapy
  Interventions: Drug: triple therapy
- Group 2: Group of ITP patients received steroids
  Interventions: Drug: Steroids
- Group 3: Normal control group

INTERVENTIONS:
Drug: triple therapy — Effect of treatment on immunity to obtain infection with hepatitis B&C
  Other Names: High dose dexamethasone together with cyclosporin and rituximab
  Groups: Group 1
Drug: Steroids — Oral or parenteral steroid therapy for ITP
  Other Names: Parenteral decadrone or oral hostacortine
  Groups: Group 2

SUMMARY:
Aim of the work To estimate frequency of viral HB & C infection in ITP patients who received triple therapy in comparison with another group treated with steroids only.

To explore risk factors and routes of transmission of viral HB & C infection in ITP patients who received triple therapy and the another group treated with steroids .

- To assess preventive measures of viral HB& C infection in the hematology ward To investigate the influence of viral HB & C infection on clinical picture, response to treatment and side effects in ITP patients who received triple therapy or steroids.

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is an autoimmune disorder characterized by isolated thrombocytopenia in the absence of other causes.ITP is mediated by antiplatelet autoantibodies. Antibody-coated platelets are phagocytosed by macrophages in the reticuloendothelial system, leading to accelerated platelet clearance. Macrophages also act as antigen-presenting cells interacting with CD8+ and CD4+ T cells that in turn stimulate antibody-producing B cells.This pathogenic loop sustains autoantibody production. T cell-mediated platelet lysis and megakaryocyte immunoinjury contribute to the diverse pathobiology of ITP.

Single-agent treatments have not been successful at inducing prolonged remission.With immunosuppressive monotherapy, ITP patients usually require prolonged treatment, leading to unpleasant and sometimes serious side effects.

Recent studies combining dexamethasone and rituximab in short courses have reported encouraging results.it is postulated that adding cyclosporine to this combination may induce a more enduring remission by also targeting T cells and thereby briefly suppressing all 3 immune cell types implicated in sustaining the pathogenic loop.

Suppressing these cells simultaneously has a risk of predisposing to serious infections.it is considered it appropriate to conduct a pilot study on a small number of patients with the aim of investigating the safety and efficacy of the triple therapy.

Infectious complications, mainly caused by the use of corticosteroids and other immunosuppressive agents, are a major cause of morbidity in patients with cITP. Moreover, infections may trigger autoimmune diseases and, at least theoretically, may be a complication of an already impaired immune system. It has been reported that children have an increased incidence of infection before diagnosis of ITP.

Hepatitis B (HBV) and C (HCV) virus infections are blood-borne viruses that pose major public health threats worldwide. The World Health Organization (WHO) report released in April 2017 on the status of hepatitis worldwide documented that 1.75 million new cases of HCV infection occurred in 2015, with about 71 million people already infected, the Eastern Mediterranean region has the highest HCV prevalence rate in the world According to WHO, in 2017 Egypt had the highest HCV prevalence rate in the world . According to the IHME in 2016, there were 4,002,706 men and 3,757,236 women with chronic HCV. HCV prevalence was estimated to be 11.9% among the general population (populations at relatively low risk of exposure to HCV, such as healthy children, blood donors, antenatal clinic attendees and pregnant women), 55.6% among populations at high risk (PWID, hemodialysis, multitransfused individuals and hemophiliacs), 14.3% among populations at intermediate risk (household contacts of HCV-infected individuals, prisoners, individuals with diabetes and healthcare workers), 56.0% among populations with liver-related conditions (acute viral hepatitis, liver cirrhosis, chronic liver disease, hepatocellular carcinoma and non-Hodgkin's lymphoma) and 35.0% among special clinical populations (dermatological manifestations, rheumatologic disorders and non-liver-related malignancies Thrombocytopenia can also complicate bleeding manifestations such as variceal bleeding. It may impede the initiation and continuation of antiviral therapy, potentially decreasing the probability of successful HCV reatment.Recent studies have evaluated the underlying mechanism of thrombocytopenia in chronic HCV infection and assessed the usefulness of several therapeutic options.

Besides hepatic complications, chronic HCV infection is also associated with several extra-hepatic manifestations including thrombocytopenia. Thrombocytopenia in chronic Hcv infection is a major problem, particularly in patients with advanced liver disease. The risk of serious bleeding with severe thrombocytopenia can prevent invasive procedures including biopsies for staging.

The pathophysiology of thrombocytopenia in patients with HCV infection is thought to be multifactorial. Besides inducing an autoimmune reaction with production of antiplatelet antibodies, the virus also causes direct bone marrow suppression with resulting thrombocytopenia , chronic HCV infection induced liver fibrosis and cirrhosis leads to portal hypertension with subsequent hypersplenism and sequestration of platelets, decreased the production of thrombopoeitin, and endothelial dysfunction, all of which can contribute to thrombocytopenia.Although uncommonly used in developed countries, interferon (IFN) and ribavirin used as part of anti-HCV therapy can also contribute to low platelet count.Hepatitis B virus (HBV) infection represents a significant global health problem, since almost one third of the worlds population has serological signs of previous or present infection, and that 240 million individuals are chronic hepatitis B surface antigen (HBsAg) carriers. Worldwide, low rates of serological HBsAg positivity (0.2%-0.5%) and signs of previous HBV contact [4%-6% HBsAg negative/anti-hepatitis B core antigen antibodies (anti-HBc)positive subjects] are registered in north western and central Europe, north America and Australia. On the contrary, the highest prevalences are reported in China, Southeast Asia and tropical Africa (chronicinfection 8%-20%, and previous exposure 70%-95%,respectively).

It is presently well known that medications such as glucocorticoids and anticancer treatments can interfere with the host immune system and blunt the control that it exerts over HBV replication, with the potential to cause viral reactivation (HBVr) in both HBsAg positive patients and individuals with serological signs of previous resolved HBV exposure. HBVr can assume various manifestations, spanning from asymptomatic hepatitis to life threatening fulminant liver failure. This risk is most common among patients undergoing treatment for hematological tumors or those receiving hematopoietic stem cell transplantation (HSCT). Nevertheless, also patients with solid tumors, immunological diseases and inflammatory bowel diseases are exposed to the risk of HBVr.The existence of an effective vaccination and a mature treatment schedule for HBV suggests that the potential for elimination of this virus as a major public health problem in Egypt exists. In a challenging economic climate, effective targeting of prevention and treatment strategies for both HBV and HCV is essential to make best use of limited resources in Egypt, however. Recent modelling work on HCV illustrates the potential power of intervention targeting in both reducing the risk of infection spread, and improving treatment outcomes, in the Egyptian context.

ELIGIBILITY:
Inclusion Criteria:

* ITP patients received triple therapy or steroids only more than 18 years old

Exclusion Criteria:

All ITP patient less than 18 years old or treated with other regimens except triple therapy or steroids.

Patients with other bleeding disorders ITP patients with known viral hepatitis B & C infection before triple therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: On patients with Idiopathic thrombocytopenic Purpura treated with triple therapy or steroids only but more than 18 years and have no other blood diseases or not known to have hepatitis B and C
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To estimate frequency of viral HB & C infection in ITP patients who received triple therapy in comparison with another group treated with steroids and risk factors affecting infection | 1 year

SECONDARY OUTCOMES:
1-To assess preventive measures of viral HB& C infection in the hematology ward 2-to asses effect of viral hepatitis b,c on clinical picture , response to treatment and side effects in ITP patients received triple therapy | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Elyamany, Prof., Study Director — Yamany1@yahoo.com; Shymaa Mohamed Nageeb, MD, Principal Investigator — Shymaanageeb1993@gmail.com

REFERENCES:
- [Background] Choi PY, Roncolato F, Badoux X, Ramanathan S, Ho SJ, Chong BH. A novel triple therapy for ITP using high-dose dexamethasone, low-dose rituximab, and cyclosporine (TT4). Blood. 2015 Jul 23;126(4):500-3. doi: 10.1182/blood-2015-03-631937. Epub 2015 May 13. PMID 25972158
- [Background] Norgaard M, Jensen AO, Engebjerg MC, Farkas DK, Thomsen RW, Cha S, Zhao S, Sorensen HT. Long-term clinical outcomes of patients with primary chronic immune thrombocytopenia: a Danish population-based cohort study. Blood. 2011 Mar 31;117(13):3514-20. doi: 10.1182/blood-2010-10-312819. Epub 2011 Jan 24. PMID 21263148
- [Background] Kramar A, Bascoul-Mollevi C. Early stopping rules in clinical trials based on sequential monitoring of serious adverse events. Med Decis Making. 2009 May-Jun;29(3):343-50. doi: 10.1177/0272989X08327332. Epub 2008 Dec 10. PMID 19073996
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Neunert C, Lim W, Crowther M, Cohen A, Solberg L Jr, Crowther MA; American Society of Hematology. The American Society of Hematology 2011 evidence-based practice guideline for immune thrombocytopenia. Blood. 2011 Apr 21;117(16):4190-207. doi: 10.1182/blood-2010-08-302984. Epub 2011 Feb 16. PMID 21325604
- [Background] Zaja F, Baccarani M, Mazza P, Bocchia M, Gugliotta L, Zaccaria A, Vianelli N, Defina M, Tieghi A, Amadori S, Campagna S, Ferrara F, Angelucci E, Usala E, Cantoni S, Visani G, Fornaro A, Rizzi R, De Stefano V, Casulli F, Battista ML, Isola M, Soldano F, Gamba E, Fanin R. Dexamethasone plus rituximab yields higher sustained response rates than dexamethasone monotherapy in adults with primary immune thrombocytopenia. Blood. 2010 Apr 8;115(14):2755-62. doi: 10.1182/blood-2009-07-229815. Epub 2010 Feb 3. PMID 20130241
- [Background] McMillan R, Wang L, Tomer A, Nichol J, Pistillo J. Suppression of in vitro megakaryocyte production by antiplatelet autoantibodies from adult patients with chronic ITP. Blood. 2004 Feb 15;103(4):1364-9. doi: 10.1182/blood-2003-08-2672. Epub 2003 Oct 23. PMID 14576051
- [Background] Gomez-Almaguer D, Tarin-Arzaga L, Moreno-Jaime B, Jaime-Perez JC, Ceballos-Lopez AA, Ruiz-Arguelles GJ, Ruiz-Delgado GJ, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Sanchez-Cardenas M. High response rate to low-dose rituximab plus high-dose dexamethasone as frontline therapy in adult patients with primary immune thrombocytopenia. Eur J Haematol. 2013 Jun;90(6):494-500. doi: 10.1111/ejh.12102. Epub 2013 Apr 2. PMID 23470153
- [Background] Bussel JB, Lee CS, Seery C, Imahiyerobo AA, Thompson MV, Catellier D, Turenne IG, Patel VL, Basciano PA, Elstrom RL, Ghanima W. Rituximab and three dexamethasone cycles provide responses similar to splenectomy in women and those with immune thrombocytopenia of less than two years duration. Haematologica. 2014 Jul;99(7):1264-71. doi: 10.3324/haematol.2013.103291. Epub 2014 Apr 18. PMID 24747949
- [Background] Gudbrandsdottir S, Birgens HS, Frederiksen H, Jensen BA, Jensen MK, Kjeldsen L, Klausen TW, Larsen H, Mourits-Andersen HT, Nielsen CH, Nielsen OJ, Plesner T, Pulczynski S, Rasmussen IH, Ronnov-Jessen D, Hasselbalch HC. Rituximab and dexamethasone vs dexamethasone monotherapy in newly diagnosed patients with primary immune thrombocytopenia. Blood. 2013 Mar 14;121(11):1976-81. doi: 10.1182/blood-2012-09-455691. Epub 2013 Jan 4. PMID 23293082
- [Background] Apostolidis J, Tsandekidi M, Kousiafes D, Pagoni M, Mitsouli C, Karmiris T, Bakiri M, Karakasis D, Harhalakis N, Nikiforakis E. Short-course corticosteroid-induced pulmonary and apparent cerebral aspergillosis in a patient with idiopathic thrombocytopenic purpura. Blood. 2001 Nov 1;98(9):2875-7. doi: 10.1182/blood.v98.9.2875a. No abstract available. PMID 11697337
- [Background] Patel VL, Mahevas M, Lee SY, Stasi R, Cunningham-Rundles S, Godeau B, Kanter J, Neufeld E, Taube T, Ramenghi U, Shenoy S, Ward MJ, Mihatov N, Patel VL, Bierling P, Lesser M, Cooper N, Bussel JB. Outcomes 5 years after response to rituximab therapy in children and adults with immune thrombocytopenia. Blood. 2012 Jun 21;119(25):5989-95. doi: 10.1182/blood-2011-11-393975. Epub 2012 May 7. PMID 22566601
- [Background] Kuwana M, Ikeda Y. The role of autoreactive T-cells in the pathogenesis of idiopathic thrombocytopenic purpura. Int J Hematol. 2005 Feb;81(2):106-12. doi: 10.1532/ijh97.04176. PMID 15765777
- [Background] Coopamah MD, Garvey MB, Freedman J, Semple JW. Cellular immune mechanisms in autoimmune thrombocytopenic purpura: An update. Transfus Med Rev. 2003 Jan;17(1):69-80. doi: 10.1053/tmrv.2003.50004. PMID 12522773
- [Background] Cines DB, Bussel JB, Liebman HA, Luning Prak ET. The ITP syndrome: pathogenic and clinical diversity. Blood. 2009 Jun 25;113(26):6511-21. doi: 10.1182/blood-2009-01-129155. Epub 2009 Apr 24. PMID 19395674
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Zaja F, Battista ML, Pirrotta MT, Palmieri S, Montagna M, Vianelli N, Marin L, Cavallin M, Bocchia M, Defina M, Ippoliti M, Ferrara F, Patriarca F, Avanzini MA, Regazzi M, Baccarani M, Isola M, Soldano F, Fanin R. Lower dose rituximab is active in adults patients with idiopathic thrombocytopenic purpura. Haematologica. 2008 Jun;93(6):930-3. doi: 10.3324/haematol.12206. Epub 2008 Apr 9. PMID 18403395
- [Result] Babudri F, Colangiuli D, Di Lorenzo PA, Farinola GM, Omar OH, Naso F. Synthesis of poly(aryleneethynylene)s bearing glucose units as substituents. Chem Commun (Camb). 2003 Jan 7;(1):130-1. doi: 10.1039/b207753a. PMID 12611000
- See also: Related Info — http://www.anzctr.org.au/